CLINICAL TRIAL: NCT00404846
Title: Effects of Hyperbaric Oxygenation Therapy on Adaptive, Aberrant and Stereotyped Behaviors in Children With Autism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Center for Autism and Related Disorders (Other)
Collaborators: The International Child Development Resource Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 906001
Record Dates: First submitted 2006-11-27; First posted 2006-11-29 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Autism
Keywords: Hyperbaric oxygenation therapy; HBOT; Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Hyperbaric Oxygenation

INTERVENTIONS:
Procedure: Hyperbaric Oxygenation Therapy

SUMMARY:
The purpose of this investigation is to evaluate the cognitive and behavioral effects of Hyperbaric Oxygenation Therapy in children who present with a diagnosis of autism and other developmental disabilities.

DETAILED DESCRIPTION:
Positive treatment effects of HBOT have been reported in a number of studies, while others have found no demonstrable effect. Studies to date have evaluated effects on a variety of conditions, and utilized diverse research methods and generally await replication. Despite its increasing usage in children with autism, and the preliminary anecdotal reports indicating positive outcome, there is a paucity of well-controlled studies of HBOT in this population, which precludes clinicians from recommending and/or implementing it as an evidence-based treatment. It is clearly important therefore, to evaluate carefully the treatment effects of HBOT using robust research designs in this population.

Hypotheses

* Hyperbaric Oxygenation Therapy will be associated with a positive effect on symptoms of autism.
* Treatment gains obtained from Hyperbaric Oxygenation Therapy will be maintained at follow-up.

Specific Aims

* Evaluate the effects of Hyperbaric Oxygenation Therapy on behavioral and cognitive symptoms of autism before, during, and after treatment.
* Determine the percentage of children with autism who respond positively to 80 HBOT treatment cycles and the extent to which they do so.
* Determine the extent to which any observed treatment effects are maintained up to three months after HBOT.

Study duration: Two weeks baseline, 10-15 week acute phase, with 1- and 3-month follow-ups.

All participants will spend one hour per session in hyperbaric oxygen chambers, for a minimum of 6 and a maximum of 10 sessions per week. A total of 80 cycles of one hour compressions must be completed within 15 weeks for all participants

Treatment Group: Pressure and Frequency

* 1.3 atmosphere absolute (ATA)
* 24% oxygen
* One session = 1 hour
* Total of 80 cycles of one hour compressions must be completed within 15 weeks.

Placebo Group: Pressure and Frequency

* Close to ambient air pressure, but the chamber needs enough pressure to inflate: 1.05 to 1.1 atmosphere absolute (ATA)
* Room Air
* One session = 1 hour
* Total of 80 cycles of one hour compressions must be completed within 15 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Autism diagnosis
* Access to CARD clinics as necessary for the study duration
* Caregiver commitment to completing 80 sessions in 10-15 weeks

Exclusion Criteria:

* Any prior treatment with HBOT
* New dietary treatment within 3 months prior to enrollment,
* New biomedical treatment within 3 weeks prior to enrollment
* Inadequate vision or hearing for the purposes of test administration
* Non-ambulatory or require more than minimum support walking
* Unstable medical disorder
* History of, or current seizure disorder
* History of, or current asthma
* History of, or current pulmonary cysts
* History of, or current emphysema
* History of, or current severe claustrophobia
* Current otitis media
* Current sinus infection
* Current upper respiratory tract infection (URTI)

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2006-11; Primary Completion 2007-09 (Actual); Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Direct Behavioral Observations
The Vineland Adaptive Behavior Scales: Expanded Edition (VABS)
Peabody Picture Vocabulary Test (PPVT)
Test of Visual-Perceptual Skills (TVPS)
The Beery-Buktenica Developmental Test of Visual-Motor Integration (VMI)
Autism Diagnostic Observation Schedule (ADOS)
The Behavior Rating Inventory of Executive Functioning (BRIEF)

SECONDARY OUTCOMES:
Aberrant Behavior Checklist
Clinical Global Impression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Bradstreet, MD, Principal Investigator — ICDRC
Locations (1):
- Center for Autism and Related Disorders, Tarzana, California, United States

REFERENCES:
- See also: Center for Autism and Related Disorders Homepage — http://www.centerforautism.com
- See also: International Child Development Resource Center Homepage — http://www.icdrc.org/